CLINICAL TRIAL: NCT03565835
Title: Abiraterone With Discontinuation of Gonadotropin-Releasing Hormone Analogues in Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin Gartrell, Principal Investigator, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-8506
Record Dates: First submitted 2018-05-29; First posted 2018-06-21 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
Keywords: abiraterone; prostate cancer; androgen deprivation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abiraterone and Prednisone without a GnRH Analogue (Experimental): Abiraterone (1000 mg daily) with Prednisone (5 mg) with Discontinuation of GnRH Analogue Injection
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone Acetate — Abiraterone Acetate with Prednisone and with Discontinuation of GnRH Analogue
Drug: Prednisone — Abiraterone Acetate with Prednisone and with Discontinuation of GnRH Analogue

SUMMARY:
The goal of this study is to find out if patients with prostate cancer being treated with the medications abiraterone and prednisone can discontinue hormone injections (examples include leuprolide, goserelin, triptorelin and degarelix). Abiraterone and prednisone are pills used to treat patients with prostate cancer. When abiraterone and prednisone are used, hormone injections are usually continued to maintain a low testosterone level in the blood. This study is being done to find out if testosterone in the blood will stay low while abiraterone and prednisone are used without continued hormone injections.

DETAILED DESCRIPTION:
Abiraterone inhibits the CYP17A enzyme, which is a critical enzyme in androgen biosynthesis. Abiraterone has regulatory approval in metastatic castration-resistant prostate cancer (mCRPC) in both chemotherapy-naïve and in the post-docetaxel setting based upon results from two randomized phase III studies. Abiraterone is also proven to extend survival in the metastatic, hormone-naïve population based on two phase III studies. Abiraterone is a castrating agent, but, other than a small first in human study, all clinical studies have been done in conjunction with gonadotropin-releasing hormone (GnRH) analogues. Maintaining castrate level of serum testosterone is critical in the treatment of metastatic prostate cancer. It is unknown if GnRH analogues must be continued to maintain castrate levels of serum testosterone in patients treated with abiraterone.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be able to provide study-specific informed consent prior to study entry
* Age ≥ 18
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Pathologically proven diagnosis of prostate adenocarcinoma
* Patients must have metastatic prostate cancer
* Patients may have mCRPC or may have metastatic castration-sensitive disease.
* Patients must be maintained on a GnRH analogue (agonist (leuprolide, goserelin, triptorelin, histrelin, deslorelin) or antagonist (degarelix))
* The patient and the investigator have decided that the next line of cancer therapy will be abiraterone plus prednisone and the initial dose of abiraterone will be 1000 mg daily. Or patients may already be on abiraterone with prednisone at a dose of 1000 mg daily along with a GnRH analogue.
* Lab values meeting the following criteria
* Total testosterone level of <50 ng/dl
* Total bilirubin < 2.0 X Upper Limit of Normal (ULN)
* Aspartate aminotransferase (AST) ≤ 3 X ULN
* Alanine aminotransferase (ALT) ≤ 3 X ULN
* Absolute Neutrophil Count > 1.5 K/mm3
* Platelets > 100 K/mm3
* Hemoglobin ≥ 9.0 g/dL
* Calculated creatinine clearance ≥ 30 mL/min

Exclusion Criteria:

* History of bilateral orchiectomy
* History of hypopituitarism
* For patients not yet started on abiraterone with prednisone, uncontrolled hypertension (systolic blood pressure >170 mm Hg or diastolic blood pressure >100 mm Hg)
* Patients must not have New York Heart Association Class III or IV heart failure at the time of screening. Patients must not have any unstable angina, myocardial infarction, or serious uncontrolled cardiac arrhythmia within 6 months prior to registration
* Any other serious illness or medical condition that the principal investigator feels would make the patient a poor candidate for this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Gartrell, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Scher HI, Sawyers CL. Biology of progressive, castration-resistant prostate cancer: directed therapies targeting the androgen-receptor signaling axis. J Clin Oncol. 2005 Nov 10;23(32):8253-61. doi: 10.1200/JCO.2005.03.4777. PMID 16278481
- [Background] Fizazi K, Tran N, Fein L, Matsubara N, Rodriguez-Antolin A, Alekseev BY, Ozguroglu M, Ye D, Feyerabend S, Protheroe A, De Porre P, Kheoh T, Park YC, Todd MB, Chi KN; LATITUDE Investigators. Abiraterone plus Prednisone in Metastatic, Castration-Sensitive Prostate Cancer. N Engl J Med. 2017 Jul 27;377(4):352-360. doi: 10.1056/NEJMoa1704174. Epub 2017 Jun 4. PMID 28578607
- [Background] James ND, de Bono JS, Spears MR, Clarke NW, Mason MD, Dearnaley DP, Ritchie AWS, Amos CL, Gilson C, Jones RJ, Matheson D, Millman R, Attard G, Chowdhury S, Cross WR, Gillessen S, Parker CC, Russell JM, Berthold DR, Brawley C, Adab F, Aung S, Birtle AJ, Bowen J, Brock S, Chakraborti P, Ferguson C, Gale J, Gray E, Hingorani M, Hoskin PJ, Lester JF, Malik ZI, McKinna F, McPhail N, Money-Kyrle J, O'Sullivan J, Parikh O, Protheroe A, Robinson A, Srihari NN, Thomas C, Wagstaff J, Wylie J, Zarkar A, Parmar MKB, Sydes MR; STAMPEDE Investigators. Abiraterone for Prostate Cancer Not Previously Treated with Hormone Therapy. N Engl J Med. 2017 Jul 27;377(4):338-351. doi: 10.1056/NEJMoa1702900. Epub 2017 Jun 3. PMID 28578639
- [Background] Barrie SE, Potter GA, Goddard PM, Haynes BP, Dowsett M, Jarman M. Pharmacology of novel steroidal inhibitors of cytochrome P450(17) alpha (17 alpha-hydroxylase/C17-20 lyase). J Steroid Biochem Mol Biol. 1994 Sep;50(5-6):267-73. doi: 10.1016/0960-0760(94)90131-7. PMID 7918112
- [Background] O'Donnell A, Judson I, Dowsett M, Raynaud F, Dearnaley D, Mason M, Harland S, Robbins A, Halbert G, Nutley B, Jarman M. Hormonal impact of the 17alpha-hydroxylase/C(17,20)-lyase inhibitor abiraterone acetate (CB7630) in patients with prostate cancer. Br J Cancer. 2004 Jun 14;90(12):2317-25. doi: 10.1038/sj.bjc.6601879. PMID 15150570
- [Background] Planas J, Celma A, Placer J, Cuadras M, Regis L, Gasanz C, Trilla E, Salvador C, Lorente D, Morote J. Hormonal response recovery after long-term androgen deprivation therapy in patients with prostate cancer. Scand J Urol. 2016 Dec;50(6):425-428. doi: 10.1080/21681805.2016.1227876. Epub 2016 Sep 14. PMID 27628623
- [Background] de Bono JS, Logothetis CJ, Molina A, Fizazi K, North S, Chu L, Chi KN, Jones RJ, Goodman OB Jr, Saad F, Staffurth JN, Mainwaring P, Harland S, Flaig TW, Hutson TE, Cheng T, Patterson H, Hainsworth JD, Ryan CJ, Sternberg CN, Ellard SL, Flechon A, Saleh M, Scholz M, Efstathiou E, Zivi A, Bianchini D, Loriot Y, Chieffo N, Kheoh T, Haqq CM, Scher HI; COU-AA-301 Investigators. Abiraterone and increased survival in metastatic prostate cancer. N Engl J Med. 2011 May 26;364(21):1995-2005. doi: 10.1056/NEJMoa1014618. PMID 21612468
- [Background] Ryan CJ, Smith MR, de Bono JS, Molina A, Logothetis CJ, de Souza P, Fizazi K, Mainwaring P, Piulats JM, Ng S, Carles J, Mulders PF, Basch E, Small EJ, Saad F, Schrijvers D, Van Poppel H, Mukherjee SD, Suttmann H, Gerritsen WR, Flaig TW, George DJ, Yu EY, Efstathiou E, Pantuck A, Winquist E, Higano CS, Taplin ME, Park Y, Kheoh T, Griffin T, Scher HI, Rathkopf DE; COU-AA-302 Investigators. Abiraterone in metastatic prostate cancer without previous chemotherapy. N Engl J Med. 2013 Jan 10;368(2):138-48. doi: 10.1056/NEJMoa1209096. Epub 2012 Dec 10. PMID 23228172
- [Background] Bong GW, Clarke HS Jr, Hancock WC, Keane TE. Serum testosterone recovery after cessation of long-term luteinizing hormone-releasing hormone agonist in patients with prostate cancer. Urology. 2008 Jun;71(6):1177-80. doi: 10.1016/j.urology.2007.09.066. Epub 2008 Feb 15. PMID 18279929
- [Background] Kaku H, Saika T, Tsushima T, Ebara S, Senoh T, Yamato T, Nasu Y, Kumon H. Time course of serum testosterone and luteinizing hormone levels after cessation of long-term luteinizing hormone-releasing hormone agonist treatment in patients with prostate cancer. Prostate. 2006 Mar 1;66(4):439-44. doi: 10.1002/pros.20341. PMID 16329145
- [Background] Scher HI, Morris MJ, Stadler WM, Higano C, Basch E, Fizazi K, Antonarakis ES, Beer TM, Carducci MA, Chi KN, Corn PG, de Bono JS, Dreicer R, George DJ, Heath EI, Hussain M, Kelly WK, Liu G, Logothetis C, Nanus D, Stein MN, Rathkopf DE, Slovin SF, Ryan CJ, Sartor O, Small EJ, Smith MR, Sternberg CN, Taplin ME, Wilding G, Nelson PS, Schwartz LH, Halabi S, Kantoff PW, Armstrong AJ; Prostate Cancer Clinical Trials Working Group 3. Trial Design and Objectives for Castration-Resistant Prostate Cancer: Updated Recommendations From the Prostate Cancer Clinical Trials Working Group 3. J Clin Oncol. 2016 Apr 20;34(12):1402-18. doi: 10.1200/JCO.2015.64.2702. Epub 2016 Feb 22. PMID 26903579

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 35 participants signed informed consent forms to participate in the study. Three participants failed to meet eligibility criteria and were excluded from the protocol and one participant opted not to participate. As a result, 31 participants were enrolled into the study.
Groups:
- Abiraterone and Prednisone Without a GnRH Analogue: Abiraterone (1000 mg daily) with Prednisone (5 mg) with Discontinuation of Gonadotropin-releasing hormone (GnRH) Analogue Injection
  Abiraterone Acetate: Abiraterone Acetate with Prednisone and with Discontinuation of GnRH Analogue
  Prednisone: Abiraterone Acetate with Prednisone and with Discontinuation of GnRH Analogue
Period: Overall Study
Arm/Group | Abiraterone and Prednisone Without a GnRH Analogue
Started | 31
Completed | 27
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Abiraterone and Prednisone Without a GnRH Analogue
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 69 [52 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/Ethnicity data was customized as all participants enrolled into the study were either Non-Hispanic Black or Hispanic/Latino.
  Participants
    non-Hispanic Black or African-American | 21
    Hispanic or Latino | 10
Region of Enrollment [Number; unit: participants]
  United States | 31
Castration-resistant disease as AAP (Abiraterone acetate plus prednisone) indication [Count of Participants; unit: Participants] — The number/percentage of participants who were diagnosed with castration-resistant disease as a condition for AAP treatment at baseline is summarized.
  Participants | 16
Duration of Androgen deprivation therapy (ADT) prior to enrollment [Mean (Full Range); unit: months] — The mean duration of ADT treatment, in months, is summarized at baseline. ADT treatment is used to suppress the levels of serum androgens including testosterone and control metastatic castration-resistant prostate cancer (mCRPC).
  months | 29.1 [3 to 204]
Duration of Abiraterone acetate plus Prednisone (AAP) prior to enrollment [Mean (Full Range); unit: months] — For participants on an existing AAP treatment regimen at baseline the mean duration of AAP treatment, in months, is summarized.
  months | 9.2 [1 to 38]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Castrate Level of Serum Testosterone
Description: The number/percentage of patients with a castrate serum testosterone level, defined as having a serum castrate concentration <50 ng/dL when Abiraterone acetate plus prednisone (AAP) is used without GnRH analogues in metastatic prostate cancer, will be determined. Results are summarized as a number/percentage of participants.
Time Frame: Approximately 24 weeks
Population: 27 of 31 patients were evaluable at ~24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone and Prednisone Without a GnRH Analogue
Number analyzed (Participants) | 27
Participants | 25

2. Secondary Outcome: Serum Testosterone (T) Levels
Description: Mean serum testosterone (T) concentrations in patients with metastatic prostate cancer treated with abiraterone acetate plus prednisone without a GnRH analogue was measured. Results have been summarized and reported in nanograms/deciliter (ng/dL) using basic descriptive statistics.
Time Frame: Baseline and 6 months, 12 months, 18 months, 24 months, and 30 months following initiation of treatment
Population: The number of patients analyzed at each timepoint is summarized in the table below.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Abiraterone and Prednisone Without a GnRH Analogue
Number analyzed (Participants) | 29
ng/dL
  Baseline | 1.52 (3.15)
  6 months: number analyzed (Participants) | 24
  6 months | 4.46 (5.1)
  12 months: number analyzed (Participants) | 21
  12 months | 7.1 (12.62)
  18 months: number analyzed (Participants) | 21
  18 months | 8.36 (8.52)
  24 months: number analyzed (Participants) | 14
  24 months | 11.07 (18.1)
  30 months: number analyzed (Participants) | 9
  30 months | 13 (20.54)

3. Secondary Outcome: Serum Luteinizing Hormone (LH) Levels
Description: Mean serum LH levels in patients with metastatic prostate cancer treated with abiraterone acetate plus prednisone without a GnRH analogue was measured. Results have been summarized and reported in International Units/Liter (IU/L) using basic descriptive statistics.
Time Frame: Baseline and 6 months, 12 months, 18 months, 24 months, and 30 months following initiation of treatment
Population: The number of patients analyzed at each timepoint is summarized in the table below.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Abiraterone and Prednisone Without a GnRH Analogue
Number analyzed (Participants) | 26
IU/L
  Baseline | 0.83 (1.17)
  6 months: number analyzed (Participants) | 24
  6 months | 17.98 (21.42)
  12 months: number analyzed (Participants) | 21
  12 months | 29.49 (26.73)
  18 months: number analyzed (Participants) | 16
  18 months | 19.32 (15.29)
  24 months: number analyzed (Participants) | 16
  24 months | 20.55 (17.27)
  30 months: number analyzed (Participants) | 10
  30 months | 21.48 (17.87)

4. Secondary Outcome: Prostate-specific Antigen (PSA) Response
Description: Mean PSA response in patients with metastatic prostate cancer treated with abiraterone acetate plus prednisone without a GnRH analogue was measured. Results have been summarized and reported in ng/mL using basic descriptive statistics.
Time Frame: Baseline and 6 months, 12 months, 18 months, 24 months, and 30 months following initiation of treatment
Population: The number of patients analyzed at each timepoint is summarized in the table below.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Abiraterone and Prednisone Without a GnRH Analogue
Number analyzed (Participants) | 28
ng/mL
  Baseline | 0.75 (1.45)
  6 Months | 0.75 (1.45)
  12 Months: number analyzed (Participants) | 19
  12 Months | 1.6 (2.35)
  18 Months: number analyzed (Participants) | 11
  18 Months | 3.2 (5.61)
  24 Months: number analyzed (Participants) | 11
  24 Months | 2.54 (3.77)
  30 Months: number analyzed (Participants) | 9
  30 Months | 2.31 (2.79)

5. Secondary Outcome: Treatment-related Adverse Events Due to Toxicity
Description: The number of patients with treatment-related adverse events due to toxicity which lead to discontinuation from the study at 24 weeks is summarized.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone and Prednisone Without a GnRH Analogue
Number analyzed (Participants) | 27
Participants | 0

6. Secondary Outcome: Radiographic Progression-free Survival (rPFS)
Description: The duration of time from trial entry until radiographic progression-free survival will be measured/reported. Progression-free survival is an assessment of the average time a patient lives without disease progression, as detected on radiographic imaging scans, or the patient dies from the disease, whichever comes first. Results have been summarized and reported in weeks using basic descriptive statistics.
Time Frame: From initiation of treatment to the end of treatment, up to approximately 41 months (~178 weeks)
Population: rPFS data was not available for 1 patient.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Abiraterone and Prednisone Without a GnRH Analogue
Number analyzed (Participants) | 30
weeks | 119 [87.1 to NA] — An upper bound 95% confidence interval was not able to be reached for rPFS due to censoring at the conclusion of the trial.

7. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is an assessment of survival from the time initiation of treatment until the time of death to death due to any cause. Results have been summarized and reported in weeks using basic descriptive statistics.
Time Frame: From initiation of treatment until the end of treatment, up to approximately 41 months
Population: OS data was not available for 1 patient.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Abiraterone and Prednisone Without a GnRH Analogue
Number analyzed (Participants) | 30
weeks | NA [102.1 to NA] — Median OS was not achieved. More than 50% of patients suppressed the censored time of 158 weeks. An upper bound 95% confidence interval was not able to be reached for OS.

8. Post Hoc Outcome: Percentage of Patients With a Castrate Serum Testosterone Level <50 ng/dL
Description: The number/percentage of patients with a castrate serum testosterone level <50 ng/dL when abiraterone acetate plus prednisone is used without GnRH analogues in metastatic prostate cancer was summarized using basic descriptive statistics.
Time Frame: 12 months, 18 months, 24 months, and 30 months following initiation of treatment
Population: The number of patients analyzed at each timepoint is summarized in the table below.
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone and Prednisone Without a GnRH Analogue
Number analyzed (Participants) | 26
Participants
  12 months | 22
  18 months: number analyzed (Participants) | 23
  18 months | 18
  24 months: number analyzed (Participants) | 22
  24 months | 16
  30 months: number analyzed (Participants) | 17
  30 months | 11

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) will be recorded from the time of consent and for at least 30 days after treatment discontinuation, up to 41 months.
Arm/Group | Abiraterone and Prednisone Without a GnRH Analogue
All-Cause Mortality (participants affected / at risk) | 3/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 16/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone and Prednisone Without a GnRH Analogue (N=31)
Fatigue (General disorders) | 1
Hot Flashes (Vascular disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 2
Prostatic Obstruction (Reproductive system and breast disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 3
Edema (General disorders) | 3
Weight Gain (Investigations) | 2
Insomnia (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-27): https://cdn.clinicaltrials.gov/large-docs/35/NCT03565835/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT03565835/ICF_001.pdf